CLINICAL TRIAL: NCT01976585
Title: A Phase I/II Study of Intratumoral Injection of rhuFlt3L/CDX-301 and Poly-ICLC in Combination With Low-Dose Radiotherapy in Low-Grade B-cell Lymphomas
Brief Title: In Situ Vaccine for Low-Grade Lymphoma: Combination of Intratumoral Flt3L and Poly-ICLC With Low-Dose Radiotherapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Joshua Brody (Other)
Collaborators: Celldex Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, Joshua Brody, Director, Lymphoma Immunotherapy Program, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 13-1347
Record Dates: First submitted 2013-10-30; First posted 2013-11-06 (Estimated); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Low-Grade B-cell Lymphoma
Keywords: Intratumoral injections; rhuFlt3L; Flt3L; CDX-301; Vaccine; Poly-ICLC; iNHL; TLR3; Low-Grade B-cell Lymphoma; Follicular; Marginal Zone; SLL; Small lymphocytic
MeSH Terms: interventions — poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rhuFlt3L/CDX-301 (Experimental): intratumoral injections on days 1-5 and 8-11. and Poly-ICLC intratumoral injection weekly, weeks 2-8
  Interventions: Drug: rhuFlt3L/CDX-301; Drug: Poly-ICLC

INTERVENTIONS:
Drug: rhuFlt3L/CDX-301 — rhuFlt3L/CDX-301 is a truncated, soluble, recombinant human fms-like tyrosine kinase-3 ligand (Flt3L), expressed in a Chinese hamster ovary cell.
  RhuFlt3L/CDX-301 is formulated as a sterile solution intended for single-use parenteral administration. Each vial contains 2.5 mg/mL rhuFlt3L/CDX-301 in a 1 mL of buffered solution composed of Sodium Phosphate and Sodium Chloride, with a pH of 7.
Drug: Poly-ICLC — Poly-ICLC is supplied by Oncovir in single-dose vials containing 1 mL of 2 mg/mL opalescent white suspension. Each milliliter of Poly-ICLC for injection contains 2 mg/mL poly-IC, 1.5 mg/mL poly-L-lysine, and 5 mg/mL sodium carboxymethylcellulose in 0.9% sodium chloride solution and adjusted to pH 7.6-7.8 with sodium hydroxide.
  Other Names: Hiltonol

SUMMARY:
Our recent trials combining local radiotherapy with intratumoral administration of TLR agonists - referred to as 'in situ vaccination' - for patients with low-grade lymphoma demonstrated safety, induction of anti-tumor CD8 T cell responses and partial and complete remissions of patients' non-irradiated sites of disease with complete remissions lasting from months to more than three years.

This iteration of the in situ vaccine approach builds on our prior work in ways that should improve its efficacy, by adding Flt3L and changing the toll-like receptors (TLR) agonist to poly-ICLC -an optimal TLR agonist for the type of dendritic cells (DC) recruited by Flt3L. The vaccine is thus in 3 phases:

1. intratumoral Flt3L administration recruits DC to the tumor
2. low-dose radiotherapy to release tumor antigens
3. intratumoral poly-ICLC administration activates tumor-antigen loaded DC

DETAILED DESCRIPTION:
Lymphomas comprise the 5th most common cancer in the U.S. with approximately 80,000 new cases diagnosed in the U.S. each year. Low-grade B-cell lymphomas are the most prevalent subtype amongst these and are considered incurable with standard therapies. Chemotherapy and monoclonal antibody therapy induce temporary remissions, though disease generally recurs, becomes progressively more resistant to therapy and ultimately therapy-resistant. Standard therapies prolong survival, though there is no standard of care regarding when to initiate therapy (versus observation) or the optimal sequence of different therapies. Novel therapies are needed with distinct mechanisms and with greater tolerability profiles. Immunotherapy has a long precedent of being able to cure low-grade lymphomas with allogeneic transplant being curative in a proportion of chemo-refractory patients, though the morbidity of this procedure reduces its broader utilization.

Previously, we completed four trials combining local radiotherapy (a standard of care for these diseases) with intratumoral administration of TLR agonists - an approach we refer to as 'in situ vaccination' for patients with previously untreated or relapsed/refractory low-grade lymphoma. We demonstrated safety, induction of anti-tumor CD8 T cell responses and partial and complete remissions of patients' non-irradiated sites of disease.1, 2 The most recent trials compared previously untreated versus relapsed/refractory patients receiving the same therapy and observed superior responses in the former group, presumably due to immunosuppressive effects of prior treatments in the latter group. The in situ vaccine is premised on pre-clinical data showing this approach to be superior to systemic TLR agonist delivery3 and our clinical results reproduce this finding; in situ vaccination yields superior response rates as compared to trials of systemic TLR agonist therapy for lymphoma.4

This iteration of the in situ vaccine approach builds on our prior work in ways that should improve its efficacy, by making two changes to the prior approach:

1. intratumoral administration of rhuFlt3L/CDX-301 to recruit dendritic cells to the tumor site
2. intratumoral administration of poly-ICLC. Flt3L has been safely administered to patients with lymphoma5 and -pre-clinically- has been shown to induce tumor leukocyte infiltration and regression of lymphoma tumors.6, 7 A total of 36 healthy volunteers and 294 cancer patients were treated including only industry-sponsored studies with the prior formulation of this agent (AMG 949) with excellent tolerability and 30 healthy volunteers were recently treated with the current formulation (CDX-301), again with excellent tolerability.

Poly-ICLC has been safely administered to patients with lymphoma8 and -pre-clinically- has been shown to induce natural killer (NK) cell cytolytic activity and regression of lymphoma tumors.9-11 Over 600 healthy volunteers and cancer patients in 17 trials have been treated with comparable doses of poly-ICLC as that used here with excellent tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-confirmed low-grade B-cell lymphoma or cutaneous T cell lymphoma; specifically, follicular grade 1, 2, or 3A, marginal zone or small lymphocytic lymphoma, or mycosis fungoides of any initial stage. Patients in cohort A must be relapsed/refractory after at least one prior systemic therapy and patients in cohort B must have had no prior systemic therapy.
* Patients must have at least one site of disease that is accessible for intratumoral injection percutaneously (e.g. inguinal, axillary, cervical, or subcutaneous).
* Tumor specimens must be available for immunological studies, either from a previous biopsy or a new biopsy obtained before the initiation Day 1 of the study.
* Patients must have measurable disease other than the injection site or biopsy site, i.e. greater than 1.5 cm bi-dimensionally on standard computed tomography imaging.
* ECOG Performance Status of 1 or better (corresponds to Karnofsky Performance Status (KPS) of ≥ 70)
* Patients must be 18 years of age or older.
* Adequate bone marrow function: WBC ≥ 2,000/μL; platelet count ≥ 75,000/mm3; ANC ≥ 1000/μL.
* Adequate renal function: serum creatinine ≤ 2.0mg/dL.
* Adequate hepatic function: bilirubin ≤ 1.5 mg/dL; SGOT/SGPT < 3 x upper limit of normal
* Required wash out periods for prior therapy (for cohort B):

  1. Topical therapy: 2 weeks
  2. Chemotherapy: 4 weeks
  3. Radiotherapy: 4 weeks
  4. Other investigational therapy: 4 weeks
  5. Rituximab: 12 weeks
* Patients of reproductive potential and their partners must agree to use an effective (> 90% reliability) form of contraception during the study and for 4 weeks following the last study drug administration.
* Women of reproductive potential must have negative urine pregnancy test.
* Life expectancy greater than 4 months.
* Able to comply with the treatment schedule.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Pre-existing autoimmune or antibody -mediated disease including: systemic lupus, erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, autoimmune thrombocytopenia, history of uveitis. Patients with controlled thyroid disease, or the presence of auto-antibodies without clinical autoimmune disease, are permitted on study.
* Known history of human immunodeficiency virus (HIV).
* Patients with active infection.
* Known CNS metastases.
* Prior malignancy (active within 5 years of screening) except basal cell or completely excised non-invasive squamous cell carcinoma of the skin, or in situ squamous cell carcinoma of the cervix.
* History of allergic reactions to compounds of similar composition to either CDX-301 or poly-ICLC.
* Current anticoagulant therapy. (ASA ≤ 325 mg per day is allowed.).
* Significant cardiovascular disease (i.e. NYHA class 3 congestive heart failure; myocardial infarction with the past 6 months; unstable angina; coronary angioplasty with the past 6 months; uncontrolled atrial or ventricular cardiac arrhythmias).
* Pregnant or lactating.
* Any other medical history, including laboratory abnormalities, deemed by the investigator to be likely to interfere with their participation in the study, or to interfere with the interpretation of the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-01-03 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
response rate | week 12
  Overall objective response rate at time of best response as defined by International Harmonization (Cheson) Criteria.

SECONDARY OUTCOMES:
safety profile | week 1
  Patient reported and clinical observation of adverse events, including changes in physical examination, peripheral blood hematology and serum chemistry
safety profile | week 2
  Patient reported and clinical observation of adverse events, including changes in physical examination, peripheral blood hematology and serum chemistry
safety profile | week 4
  Patient reported and clinical observation of adverse events, including changes in physical examination, peripheral blood hematology and serum chemistry
safety profile | week 6
  Patient reported and clinical observation of adverse events, including changes in physical examination, peripheral blood hematology and serum chemistry
safety profile | week 8
  Patient reported and clinical observation of adverse events, including changes in physical examination, peripheral blood hematology and serum chemistry
safety profile | week 12
  Patient reported and clinical observation of adverse events, including changes in physical examination, peripheral blood hematology and serum chemistry
tumor-specific immune response | baseline
  Pre- to post-treatment induction of systemic (peripheral blood) tumor-specific immune response.
tumor-specific immune response | week 2
  Pre- to post-treatment induction of systemic (peripheral blood) tumor-specific immune response.
tumor-specific immune response | week 4
  Pre- to post-treatment induction of systemic (peripheral blood) tumor-specific immune response.
tumor-specific immune response | week 6
  Pre- to post-treatment induction of systemic (peripheral blood) tumor-specific immune response.
tumor-specific immune response | week 8
  Pre- to post-treatment induction of systemic (peripheral blood) tumor-specific immune response.
tumor-specific immune response | week 12
  Pre- to post-treatment induction of systemic (peripheral blood) tumor-specific immune response.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Brody, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] Brody JD, Ai WZ, Czerwinski DK, Torchia JA, Levy M, Advani RH, Kim YH, Hoppe RT, Knox SJ, Shin LK, Wapnir I, Tibshirani RJ, Levy R. In situ vaccination with a TLR9 agonist induces systemic lymphoma regression: a phase I/II study. J Clin Oncol. 2010 Oct 1;28(28):4324-32. doi: 10.1200/JCO.2010.28.9793. Epub 2010 Aug 9. PMID 20697067
- [Background] Kim YH, Gratzinger D, Harrison C, Brody JD, Czerwinski DK, Ai WZ, Morales A, Abdulla F, Xing L, Navi D, Tibshirani RJ, Advani RH, Lingala B, Shah S, Hoppe RT, Levy R. In situ vaccination against mycosis fungoides by intratumoral injection of a TLR9 agonist combined with radiation: a phase 1/2 study. Blood. 2012 Jan 12;119(2):355-63. doi: 10.1182/blood-2011-05-355222. Epub 2011 Nov 1. PMID 22045986
- [Background] Li J, Song W, Czerwinski DK, Varghese B, Uematsu S, Akira S, Krieg AM, Levy R. Lymphoma immunotherapy with CpG oligodeoxynucleotides requires TLR9 either in the host or in the tumor itself. J Immunol. 2007 Aug 15;179(4):2493-500. doi: 10.4049/jimmunol.179.4.2493. PMID 17675511
- [Background] Link BK, Ballas ZK, Weisdorf D, Wooldridge JE, Bossler AD, Shannon M, Rasmussen WL, Krieg AM, Weiner GJ. Oligodeoxynucleotide CpG 7909 delivered as intravenous infusion demonstrates immunologic modulation in patients with previously treated non-Hodgkin lymphoma. J Immunother. 2006 Sep-Oct;29(5):558-68. doi: 10.1097/01.cji.0000211304.60126.8f. PMID 16971811
- [Background] Chen W, Chan AS, Dawson AJ, Liang X, Blazar BR, Miller JS. FLT3 ligand administration after hematopoietic cell transplantation increases circulating dendritic cell precursors that can be activated by CpG oligodeoxynucleotides to enhance T-cell and natural killer cell function. Biol Blood Marrow Transplant. 2005 Jan;11(1):23-34. doi: 10.1016/j.bbmt.2004.08.004. PMID 15625541
- [Background] Zhang YL, Wei YJ, Deng YC, Wang YD, Liu CZ, Su L, Yang KG, Chen SS. Human Flt3 ligand from Pichia pastoris inhibits growth of lymphoma and colon adenocarcinoma in mice. J Exp Ther Oncol. 2006;5(3):161-6. PMID 16528967
- [Background] Esche C, Subbotin VM, Maliszewski C, Lotze MT, Shurin MR. FLT3 ligand administration inhibits tumor growth in murine melanoma and lymphoma. Cancer Res. 1998 Feb 1;58(3):380-3. PMID 9458075
- [Background] Giantonio BJ, Hochster H, Blum R, Wiernik PH, Hudes GR, Kirkwood J, Trump D, Oken MM. Toxicity and response evaluation of the interferon inducer poly ICLC administered at low dose in advanced renal carcinoma and relapsed or refractory lymphoma: a report of two clinical trials of the Eastern Cooperative Oncology Group. Invest New Drugs. 2001;19(1):89-92. doi: 10.1023/a:1006458232384. PMID 11291838
- [Background] Black PL, Hartmann D, Pennington R, Phillips H, Schneider M, Tribble HR, Talmadge JE. Effect of tumor burden and route of administration on the immunotherapeutic properties of polyinosinic-polycytidylic acid stabilized with poly-L-lysine in carboxymethyl cellulose [Poly(I,C)-LC]. Int J Immunopharmacol. 1992 Nov;14(8):1341-53. doi: 10.1016/0192-0561(92)90005-6. PMID 1464467
- [Background] Storch E, Kirchner H, Schirrmacher V. Prolongation of survival of mice bearing the Eb and ESb lymphoma by treatment with interferon inducers alone or in combination with Corynebacterium parvum. Cancer Immunol Immunother. 1986;23(3):179-84. doi: 10.1007/BF00205647. PMID 2431778
- [Background] Fresa KL, Korngold R, Murasko DM. Induction of natural killer cell activity of thoracic duct lymphocytes by polyinosinic-polycytidylic acid (poly(I:C)) or interferon. Cell Immunol. 1985 Apr 1;91(2):336-43. doi: 10.1016/0008-8749(85)90231-x. PMID 2581698